CLINICAL TRIAL: NCT04711122
Title: The Role of Prophylactic Antibiotics in Prevention of Spontaneous Bacterial Peritonitis in Compensated Liver Cirrhosis With Upper Gastrointestinal Bleeding
Brief Title: Prophylactic Antibiotics in Prevention of Spontaneous Bacterial Peritonitis in Compensated Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nariman Gamal Abd Elhakeem, Principal investigator, Assiut University
Other Study IDs: 12345678
Record Dates: First submitted 2020-03-25; First posted 2021-01-15 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Liver Cirrhosis; Upper Gastrointestinal Bleeding
Keywords: Liver cirrhosis; Childscore A
MeSH Terms: conditions — Liver Cirrhosis; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Role of prophylactic antibiotics in childscore A: Role of prophylaxis against infections in progression of cirrhotic patients with childscore A
  Interventions: Drug: Third generation cephalosporin antibiotics

INTERVENTIONS:
Drug: Third generation cephalosporin antibiotics — Assessment of antibiotic effect

SUMMARY:
timely short-term antibiotic prophylaxis is an essential step in the management of these patients . Prophylaxis must be instituted as early as variceal hemorrhage is suspected, and timely administration has been associated with a reduced re-bleeding rate and lower mortality .

More recently, the American Association for the Study of Liver Diseases (AASLD), the Department of Veterans Affairs (VA), and the American Society for Gastrointestinal Endoscopy (ASGE) recommended antibiotic prophylaxis in all cirrhotic patients with UGIB, regardless of its source (i.e. variceal or non-variceal) or the presence of ascites.

DETAILED DESCRIPTION:
cute variceal bleeding is one of the major causes of death in cirrhotic patients . It is also the major cause of upper gastrointestinal (GI) bleeding in cirrhotic patients, accounting for 70% of cases . Mortality during the first episode is estimated to 15-20% but is higher in severe patients (Child Pugh C), at around 30%, whereas it is very low in patients with compensated cirrhosis (Child Pugh A).

Hemorrhage from gastro-esophageal varices is a devastating complication of portal hypertension. Although the in-hospital mortality of acute variceal bleeding was up to 40% about 20 years ago, it was decreased to about 15-20% in recent years.20 One of the main reasons in the decrease of mortality has been ascribed to the alertness of clinicians in the treatment and prophylaxis of associated bacterial infections. The prevalence of bacterial infections in cirrhotic patients with gastrointestinal hemorrhage has been up to 52%-66%.

Therefore, timely short-term antibiotic prophylaxis is an essential step in the management of these patients. Prophylaxis must be instituted as early as variceal hemorrhage is suspected, and timely administration has been associated with a reduced re-bleeding rate and lower mortality .

More recently, the American Association for the Study of Liver Diseases (AASLD), the Department of Veterans Affairs (VA), and the American Society for Gastrointestinal Endoscopy (ASGE) recommended antibiotic prophylaxis in all cirrhotic patients with UGIB, regardless of its source (i.e. variceal or non-variceal) or the presence of ascites.

The importance of prophylaxis is incontrovertible in patients with advanced cirrhosis, whereas in patients with less severe disease, conflicting data have been published. In a retrospective study, Child A patients had a low rate of bacterial infection (2%) in the absence of antibiotic prophylaxis, and there was no difference in mortality between patients on and off antibiotics .

In contrast, antibiotics were associated with a marked mortality reduction in Child C patients. However, more prospective studies are needed to assess whether antibiotic prophylaxis can be avoided in Child A patients .

Thus, this study will be conducted to investigate the necessity of prophylactic antibiotic in compensated cirrhotic patients with UGIB and to evaluate its influence on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child score "A" Cirrhotic patients
* Hematemesis and / or melena.

Exclusion Criteria:

* Patient with unsuccessful endoscopic hemostasis
* Patients who already have signs of infections (elevation in the body temperature, elevation in white blood cells above 10,000 cell/mmᵌ);
* Patients with occult infection (defined as positive blood cultures obtained before antibiotic prophylaxis)
* Patients using antibiotics before endoscopy.
* Patients refuse to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cirrhotic patients with childscore A
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Prophylactic antibiotics in cirrhotic patients. | 1 year
  Rate of infection in patients using prophylactic antibiotics in Child A cirrhotic patients presented with upper gastrointestinal bleeding according to blood culture and chest x ray.

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Gamal, MD, Principal Investigator — Assiut University

REFERENCES:
- See also: Related Info — https://doi.org/10.1002/hep.1840050320